CLINICAL TRIAL: NCT00840177
Title: S0919, A Phase II Study of Idarubicin and Ara-C in Combination With Pravastatin for Poor-Risk Acute Myelogenous Leukemia
Brief Title: S0919 Idarubicin, Cytarabine, and Pravastatin in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0919; S0919 (Other: SWOG); U10CA032102 (NIH); NCI-2009-01183 (Other: NCI)
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Cytarabine; Idarubicin; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): Induction (1 cycle):
  pravastatin 1280 mg/d PO D 1-8 idarubicin 12 mg/m2/d IV D 4-6 cytarabine 1.5 g/m2/d continuous IV D 4-7
  Consolidation (up to 2 cycles):
  pravastatin 1280 mg/d PO D 1-6 idarubicin 12 mg/m2/d IV D 4-5 cytarabine 1.5 g/m2/d continuous IV D 4-5
  Interventions: Drug: cytarabine; Drug: idarubicin; Drug: pravastatin sodium

INTERVENTIONS:
Drug: cytarabine — 1.5 g/m2/day given by continuous IV on days 4-7
Drug: idarubicin — 12 mg/m2/day given intravenously over 10-15 minutes on days 4-6
Drug: pravastatin sodium — 1,280 mg/day given orally on days 1-8

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Pravastatin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Pravastatin may also help idarubicin and cytarabine work better by making cancer cells more sensitive to the drugs. Giving idarubicin and cytarabine together with pravastatin may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving idarubicin and cytarabine together with pravastatin works in treating patients with relapsed acute myeloid leukemia (AML).

ADDITIONAL BACKGROUND: S0919 was initially designed for patients with relapsed acute myeloid leukemia (AML), where the patient's preceding remission had lasted ≥ 3 months. The null response rate was 30%. The study closed to accrual on Nov 1, 2012 after meeting the defined criterion for a positive study; and the results are being submitted to the American Society of Clinical Oncology meeting. Based on the promising results from this trial, the trial has now been amended to evaluate this therapeutic regimen in poor-risk patients (patients with newly diagnosed acute myeloid leukemia (AML) arising out of myelodysplastic syndrome (MDS), primary refractory acute myeloid leukemia (AML), and relapsed acute myeloid leukemia (AML) with the patient's preceding remission lasting < 6 months).

DETAILED DESCRIPTION:
COHORTS:

Cohort 1 (Initial cohort: Relapsed AML with previous remission ≥ 3 months), Cohort 2 (Poor-risk cohort: MDS transformed to AML), Cohort 3 (Poor-risk cohort: Refractory or relapsed AML with previous remission < 6 months)

OBJECTIVES:

* To test whether the complete remission (CR) rate (including CR with incomplete recovery) in patients with relapsed acute myeloid leukemia (AML) treated with idarubicin and cytarabine in combination with pravastatin is sufficiently high to warrant a phase III investigation.
* To estimate relapse-free survival and overall survival rates in these patients.
* To estimate the frequency and severity of toxicities of this regimen in these patients.
* To evaluate, in a preliminary manner, whether pre-study cytogenetic features correlate with response in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive oral pravastatin once daily on days 1-8, idarubicin IV over 10-15 minutes on days 4-6, and cytarabine IV continuously on days 4-7. Patients achieving complete remission proceed to consolidation therapy.
* Consolidation therapy: Beginning 30-60 days after the start of induction therapy, patients receive oral pravastatin once daily on days 1-6 and idarubicin IV over 10-15 minutes and cytarabine IV continuously on days 4 and 5. Treatment repeats approximately every 5 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Cohort 1 (Initial cohort: Relapsed AML with previous remission >/= 3 months) is permanently closed to accrual DISEASE CHARACTERISTICS

* Patients must have a previous morphologically confirmed diagnosis of acute myeloid leukemia (AML). Note: This protocol uses the World Health Organization (WHO) diagnostic criteria for acute myeloid leukemia (AML) (see Section 4.1). Patients with acute promyelocytic leukemia (APL, FAB, M3) or blastic transformation of chronic myelogenous leukemia (CMML) are not eligible.
* Patients must have received at least one prior chemotherapy regimen for their acute myeloid leukemia (AML) and they may have received any type of chemotherapy. They must have achieved complete remission (CR), lasting at least three months with their last induction regimen and they must have relapsed after the last regimen. Relapse must be documented by a bone marrow examination demonstrating > 5% blasts in the bone marrow not attributable to another cause. Refractory patients and patients who have received autologous or allogeneic stem cell transplantation are not eligible. Administration of hydroxyurea to control high white blood cell (WBC) count prior to, during and after registration is permitted.
* Patients must not have symptomatic congestive heart failure, coronary artery disease, cardiomyopathy, or uncontrolled arrhythmias. Either an echocardiogram or multiple-gated acquisition (MUGA) scan with an ejection fraction ≥ 45% must be obtained within 28 days prior to registration. (Either method for measuring cardiac function is acceptable, however, the same scan must be used throughout treatment and follow-up to monitor the patient for cardiac toxicity.) If patient has symptoms suggestive of ischemia or congestive heart failure after that cardiac evaluation was done, a repeat study must be obtained prior to registration.
* Patients must have a serum creatinine < 2.0 mg/dl within 14 days prior to registration.
* Patients must have a total bilirubin ≤ 2.0 x Institutional Upper Limit of Normal (IULN) within 14 days prior to registration, unless the elevation is due primarily to elevated unconjugated hyperbilirubinemia secondary to Gilbert's syndrome or hemolysis and not to liver dysfunction.
* Patients must have SGOT (AST) ≤ 3.0 x IULN and SGPT (ALT) ≤ 3.0 x IULN within 14 days prior to registration. Treatment may begin with SGOT/SGPT above those limits, if the abnormalities are thought to be due to the patient's leukemia.
* Patients must have Zubrod performance status of 0-2 (see Section 10.8).
* Patients must be ≥ 18 years of age.
* Patients must not have clinical evidence of leptomeningeal disease (a spinal tap does not need to be performed).
* Patients not known to be HIV+ must be tested for HIV infection (the human immunodeficiency virus) within 14 days prior to registration (see Section 2.0 for justification). Patients who are HIV+ may be eligible providing they meet all of the following additional criteria within 14 days prior to registration:

  1. Patient must have no history of AIDS defining events.
  2. CD4 cells ≥ 500/mm3.
  3. Viral load of < 50 copies HIV mRNA/mm3 if on cART or < 25,000 copies HIV mRNA if not on cART.
  4. No zidovudine or stavudine as part of cART. Patients who are HIV+ and do not meet all of these criteria will not be eligible for this study.
* Patients with prior malignancy (other than AML) are eligible. However, the patient must be in remission from the prior malignancy and have completed all chemotherapy and radiotherapy at least 6 months prior to registration and all treatment related toxicities must have been resolved. NOTE: For patients with prior history of malignancy who have received anthracyclines or mediastinal/pericardial radiation in the past, the risk versus benefit of therapy should be weighed, particularly in the setting of receiving consolidation therapy.
* Patients must not have a systemic fungal, bacterial, viral or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Southwest Oncology Group patients must be registered on SWOG-9007 ("Cytogenetic Studies in Leukemia Patients"). Collection of pretreatment marrow specimens must be completed within 28 days prior to registration. Pretreatment specimens of bone marrow (or peripheral blood if the marrow aspirate is a dry tap) must be submitted to an approved Southwest Oncology Group Cytogenetics Laboratory for cytogenetics analysis. Note that protocol SWOG-9007 also requires submission of specimens at additional timepoints.
* Southwest Oncology Group patients must be offered participation in S9910 ("Leukemia Centralized Reference Laboratories and Tissue Repositories Ancillary"). If consent is given, collection of pretreatment blood and/or marrow specimens must be completed within 28 days prior to registration. If the patient consents to participate in S9910, pretreatment specimens of marrow and/or peripheral blood must be submitted to the Southwest Oncology Group Myeloid Repository at the University of New Mexico for cellular and molecular studies. Note that protocol S9910 also requests submission of specimens at additional timepoints.
* Women of reproductive potential must have a negative pregnancy test within 14 days prior to registration. Patients must not be pregnant or nursing because of the teratogenic potential of the drugs used in this study. Women/men of reproductive potential must have agreed to use an effective contraceptive method.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base.

Cohort 2 (MDS transformed to AML) is permanently closed to accrual AND Cohort 3 (relapsed/refractory AML) is permanently closed to accrual

DISEASE CHARACTERISTICS:

* For patients registered to relapsed/refractory (Cohort 3), morphologically confirmed diagnosis of acute myeloid leukemia (AML)
* Patient registered to the myelodysplastic syndrome (MDS) transformed to acute myeloid leukemia (AML) cohort (Cohort 2) patients must have a previous morphologically confirmed diagnosis of myelodysplastic syndrome/chronic myelomonocytic leukemia (MDS/CMML). Patients may have received previous non-intensive therapy (such as: azacitidine, decitabine, low-dose cytarabine, lenalidomide) given treatment of myelodysplastic syndrome/chronic myelomonocytic leukemia (MDS/CMML) (with up to 20% blasts). At time of registration, patient must have morphologically confirmed diagnosis of acute myeloid leukemia (AML).
* Patients with acute promyelocytic leukemia (i.e., APL, FAB M3) or blastic transformation of chronic myelogenous leukemia are not eligible
* Patients must not have received autologous or allogeneic stem cell transplant.
* Patients in the relapsed/refractory acute myeloid leukemia (AML) cohort (Cohort 3) must:

  * Have received ≥ 1 prior chemotherapy regimen for acute myeloid leukemia (AML)

    * Any type of prior chemotherapy allowed
    * Administration of hydroxyurea to control high white blood cell (WBC) prior to, during, and after registration is permitted
  * Relapse must be documented by a bone marrow examination demonstrating > 5% blasts in the bone marrow not attributable to another cause
  * Patient must not have received chemo within 14 days prior to registration
* Primary refractory patients eligible if, on Day 14 of previous chemo regimen, they have significant residual disease. Patients who received only hypomethylating agent or low dose therapy for Induction are not considered primary refractory for this study and are not eligible.
* Relapsed patients must have achieved a complete remission (CR) or CR with incomplete blood count recovery that lasted < 6 months after the last induction regimen
* No clinical evidence of leptomeningeal disease
* Pretreatment (collected within 28 days of registration) cytogenetics must be performed on all patients.
* Patients must have complete history and physical exam within 28 days prior to registration.

PATIENT CHARACTERISTICS:

* No symptomatic congestive heart failure, coronary artery disease, cardiomyopathy, or uncontrolled arrhythmias

  * Ejection fraction ≥ 45% by echocardiogram or MUGA scan within 28 days prior to registration (or within 14 days prior to registration if the patient has received anthracycline in the 28 day window)
* Zubrod performance status 0-2
* Serum creatinine ≤ 2.0 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 times ULN (unless elevation is primarily due to elevated unconjugated hyperbilirubinemia secondary to Gilbert's syndrome or hemolysis AND not due to liver dysfunction)
* AST and ALT ≤ 3.0 times ULN
* Not pregnant or nursing and negative pregnancy test within 14 days prior to registration. Females of child-bearing potential must agree to use effective contraception
* No HIV positivity unless the following criteria are met:

  * No history of AIDS-defining events
  * CD4 count ≥ 500/mm³
  * Viral load < 25,000 copies (< 50 copies if on combination antiretroviral therapy)
  * Not receiving zidovudine or stavudine as part of combination antiretroviral therapy
* No uncontrolled systemic fungal, bacterial, viral, or other infection, defined as exhibiting ongoing signs/symptoms related to the infection with no improvement despite appropriate antibiotics or other treatment
* Patients with prior malignancy (other than AML and MDS/CMML) eligible provided patient is in remission from that malignancy at least 6 months prior to registration. Except for acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) treatment, all treatment related toxicities must have been resolved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-12-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Study Chair — The Cleveland Clinic
Locations (185):
- United States (185):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford Cancer Institute, Palo Alto, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Memorial and Saint Elizabeth's Health Care Services LLP, Swansea, Illinois
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton Health Center, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Hematology Oncology Associates East PC, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Statler A, Othus M, Erba HP, Chauncey TR, Radich JP, Coutre S, Advani A, Nand S, Ravandi F, Mukherjee S, Sekeres MA. Comparable outcomes of patients eligible vs ineligible for SWOG leukemia studies. Blood. 2018 Jun 21;131(25):2782-2788. doi: 10.1182/blood-2018-01-826693. Epub 2018 Apr 4. PMID 29618479

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Month: Participants with previous morphologically confirmed acute myeloid leukemia (AML), and preceding remission lasting ≥ 3 months
- Poor-risk Cohort: MDS Transformed to AML: Participants with acute myeloid leukemia (AML) who had a previous morphologically confirmed diagnosis of myelodysplastic syndrome(MDS)/Chronic Myelomonocytic Leukemia (CMML) and for which they may have received previous non-intensive therapy.
- Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission: Participants with previous morphologically confirmed acute myeloid leukemia (AML), and preceding remission lasting < 6 months.
Period: Overall Study
Arm/Group | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Month | Poor-risk Cohort: MDS Transformed to AML | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission
Started | 36 | 29 | 50
Treated | 36 | 29 | 46
Assessed for AEs | 35 | 29 | 46
Completed | 18 | 20 | 39
Not Completed | 18 | 9 | 11
Not completed — Adverse Event | 5 | 1 | 1
Not completed — Refusal unrelated to adverse events | 1 | 0 | 1
Not completed — Progression/relapse | 2 | 0 | 0
Not completed — Death | 4 | 5 | 5
Not completed — not protocol specified | 6 | 3 | 0
Not completed — Ineligible | 0 | 0 | 3
Not completed — Did not start treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who started treatment
Groups:
- Poor-risk Cohort: MDS Transformed to AML: Participants with acute myeloid leukemia (AML) who had a previous morphologically confirmed diagnosis of MDS/CMML and for which they may have received previous non-intensive therapy.
- Total: Total of all reporting groups
Arm/Group | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Month | Poor-risk Cohort: MDS Transformed to AML | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission | Total
Number analyzed (Participants) | 36 | 29 | 46 | 111
Age, Continuous [Median (Full Range); unit: years] | 58.6 [23.2 to 78.2] | 64.9 [21.8 to 77.1] | 57.3 [23.1 to 74.9] | 60.7 [21.8 to 78.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 22 | 54
  Male | 17 | 16 | 24 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 4 | 9
  Not Hispanic or Latino | 29 | 28 | 38 | 95
  Unknown or Not Reported | 2 | 1 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 1 | 2 | 6
  White | 30 | 28 | 35 | 93
  More than one race | 0 | 0 | 3 | 3
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate (Including CR With Incomplete Recovery)
Description: Participants who achieved morphological complete remission with or without incomplete blood count recovery.
  Per the Revised Recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia, morphologic complete remission requires that the patient achieve the morphologic leukemia-free state and have an absolute neutrophil count of more than 1,000/μL and platelets of ≥ 100,000/μL.
Time Frame: Up to 5 years after registration
Population: Eligible participants who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Month | Poor-risk Cohort: MDS Transformed to AML | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission
Number analyzed (Participants) | 36 | 29 | 46
Participants | 27 | 14 | 14

2. Secondary Outcome: Frequency and Severity of Toxicity as Assessed by NCI CTCAE Version 3.0
Description: Number of patients with Grade 3-5 adverse events that were possibly, probably or definitely related to study drug are reported by given type of adverse event
Time Frame: Up to 5 years post registration
Population: Eligible patients who were assessed for adverse events
Measure: Number; unit: Participants
Arm/Group | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Month | Poor-risk Cohort: MDS Transformed to AML | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission
Number analyzed (Participants) | 35 | 29 | 46
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 2 | 2
  AST, SGOT | 0 | 3 | 1
  Acidosis (metabolic or respiratory) | 0 | 1 | 0
  Albumin, serum-low (hypoalbuminemia) | 1 | 3 | 6
  Alkaline phosphatase | 0 | 0 | 1
  Alkalosis (metabolic or respiratory) | 0 | 1 | 0
  Anorexia | 1 | 1 | 0
  Bilirubin (hyperbilirubinemia) | 2 | 2 | 0
  Blood/Bone Marrow-Other (Specify) | 2 | 1 | 0
  Bone marrow cellularity | 1 | 0 | 0
  Calcium, serum-low (hypocalcemia) | 2 | 5 | 3
  Carbon monoxide diffusion capacity (DL(co)) | 1 | 4 | 1
  Cardiac General-Other (Specify) | 1 | 0 | 0
  Cardiac-ischemia/infarction | 0 | 1 | 0
  Colitis, infectious (e.g., Clostridium difficile) | 0 | 1 | 1
  Conduction abnormality - Asystole | 1 | 0 | 0
  Confusion | 1 | 0 | 0
  Constitutional Symptoms-Other (Specify) | 0 | 2 | 0
  Creatinine | 0 | 3 | 2
  Diarrhea | 3 | 4 | 8
  Distention/bloating, abdominal | 0 | 2 | 0
  Dry mouth/salivary gland (xerostomia) | 0 | 1 | 0
  Dyspnea (shortness of breath) | 2 | 1 | 2
  Edema: limb | 0 | 2 | 0
  Esophagitis | 1 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 3 | 2 | 2
  Febrile neutropenia | 20 | 18 | 32
  Glucose, serum-high (hyperglycemia) | 1 | 2 | 0
  Hemoglobin | 11 | 14 | 21
  Hemorrhage, GI - Duodenum | 0 | 1 | 0
  Hemorrhage, GU - Vagina | 1 | 0 | 0
  Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS | 0 | 0 | 1
  Hemorrhage, pulmonary/upper respiratory - Nose | 0 | 0 | 1
  Hemorrhage/Bleeding-Other (Specify) | 1 | 0 | 0
  Hypertension | 1 | 0 | 0
  Hypotension | 1 | 2 | 1
  Hypoxia | 1 | 2 | 3
  Ileus, GI (functional obstruction of bowel) | 1 | 2 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 4 | 4 | 7
  Inf (clin/microbio) w/Gr 3-4 neuts - Bronchus | 1 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Kidney | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 5 | 2 | 6
  Inf (clin/microbio) w/Gr 3-4 neuts - Meninges | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Sinus | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 0 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Small bowel | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Stomach | 0 | 0 | 1
  Infection with unknown ANC - Blood | 1 | 2 | 4
  Infection with unknown ANC - Lung (pneumonia) | 0 | 1 | 0
  Infection with unknown ANC - Mucosa | 0 | 0 | 1
  Infection with unknown ANC - Sinus | 1 | 0 | 0
  Infection with unknown ANC - Small bowel NOS | 0 | 1 | 0
  Infection-Other (Specify) | 1 | 1 | 0
  Left ventricular diastolic dysfunction | 2 | 0 | 0
  Leukocytes (total WBC) | 16 | 11 | 17
  Lipase | 1 | 0 | 0
  Lymphopenia | 6 | 5 | 9
  Magnesium, serum-high (hypermagnesemia) | 0 | 1 | 0
  Mental status | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 0 | 0 | 1
  Mucositis/stomatitis (clinical exam) - Pharynx | 0 | 0 | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 1 | 0 | 1
  Musculoskeletal/Soft Tissue-Other (Specify) | 0 | 1 | 0
  Nausea | 2 | 1 | 3
  Necrosis, GI - Small bowel NOS | 0 | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 14 | 15 | 16
  Obstruction, GI - Small bowel NOS | 0 | 1 | 0
  Ocular/Visual-Other (Specify) | 1 | 0 | 0
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 0 | 0 | 2
  Pain - Abdomen NOS | 1 | 3 | 0
  Pain - Bone | 0 | 0 | 1
  Pain - Esophagus | 0 | 0 | 1
  Pain - Extremity-limb | 0 | 0 | 1
  Pain - Oral cavity | 0 | 0 | 3
  Pain - Peritoneum | 0 | 1 | 0
  Phosphate, serum-low (hypophosphatemia) | 2 | 4 | 2
  Platelets | 17 | 16 | 19
  Pleural effusion (non-malignant) | 0 | 1 | 0
  Potassium, serum-high (hyperkalemia) | 0 | 2 | 0
  Potassium, serum-low (hypokalemia) | 6 | 3 | 3
  Pulmonary hypertension | 1 | 0 | 0
  Pulmonary/Upper Respiratory-Other (Specify) | 0 | 1 | 0
  Rash/desquamation | 0 | 0 | 1
  Renal failure | 0 | 0 | 2
  Renal/Genitourinary-Other (Specify) | 0 | 1 | 0
  SVT and nodal arrhythmia - Atrial fibrillation | 1 | 1 | 0
  SVT and nodal arrhythmia - Atrial flutter | 1 | 0 | 0
  Sodium, serum-high (hypernatremia) | 1 | 0 | 0
  Sodium, serum-low (hyponatremia) | 1 | 0 | 1
  Syncope (fainting) | 1 | 0 | 0
  Typhlitis (cecal inflammation) | 0 | 0 | 1
  Ulcer, GI - Duodenum | 0 | 1 | 0
  Ulceration | 0 | 0 | 1
  Vomiting | 2 | 2 | 0
  Weight loss | 0 | 0 | 2

3. Other Pre Specified Outcome: Correlation Between Pre-study Cytogenetic Features and Response
Time Frame: 5 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS is calculated for all participants from the date of initial registration on study until death from any cause. Observations for participants last known to be alive were censored.
Time Frame: OS assessed for up to 5 years, median OS reported
Population: Eligible participants who started treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Month | Poor-risk Cohort: MDS Transformed to AML | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission
Number analyzed (Participants) | 36 | 29 | 46
months | 10 [7 to 12] | 10 [4 to 18] | 4 [3 to 6]

5. Other Pre Specified Outcome: Relapse-free Survival (RFS)
Description: RFS is calculated for participants who have achieved a complete response (CR) or CR with incomplete blood count recovery (CRi). RFS will be measured from the date of CR or CRi until relapse from CR or CRi for death from any cause. Observation is censored at the date of last follow-up for patients last known to be alive without report of relapse.
  Per the Revised Recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia, morphologic complete remission requires that the patient achieve the morphologic leukemia-free state and have an absolute neutrophil count of more than 1,000/μL and platelets of ≥ 100,000/μL.
Time Frame: RFS assessed for up to 5 years, median RFS reported
Population: Eligible participants who started treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Month | Poor-risk Cohort: MDS Transformed to AML | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission
Number analyzed (Participants) | 36 | 29 | 46
months | 9 [5 to 20] | 19.4 [4.3 to NA] — The upper 95% confidence limit for the median cannot be estimated using the method of Brookmeyer and Crowley (1982). | 2.7 [0.3 to 18.9]

ADVERSE EVENTS:
Time Frame: Up to 5 years post registration
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. All adverse events, regardless of attribution or grade, are reported for patients who received study treatment. 1 patient in the initial cohort was taken off protocol therapy before AEs were assessed.
Groups:
- Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Mnths: Participants with previous morphologically confirmed acute myeloid leukemia (AML), and preceding remission lasting ≥ 3 months
Arm/Group | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Mnths | Poor-risk Cohort: MDS Transformed to AML | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission
All-Cause Mortality (participants affected / at risk) | 27/36 | 20/29 | 41/46
Serious Adverse Events (participants affected / at risk) | 5/35 | 8/29 | 10/46
Other Adverse Events (participants affected / at risk) | 34/35 | 28/29 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Mnths (N=35) | Poor-risk Cohort: MDS Transformed to AML (N=29) | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac General-Other (Cardiac disorders) | 1 | 1 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 0 | 1 | 0
Conduction abnormality - Asystole (Cardiac disorders) | 1 | 0 | 0
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 1 | 0 | 0
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 0 | 3
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 0 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1 | 0 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 1 | 2 | 5
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 0 | 1 | 0
Infection with unknown ANC - Small bowel NOS (Infections and infestations) | 0 | 1 | 0
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 1 | 4 | 1
Lymphopenia (Investigations) | 1 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 0 | 0
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hemorrhage, CNS (Nervous system disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Cohort: Relapsed AML With Previous Remission ≥ 3 Mnths (N=35) | Poor-risk Cohort: MDS Transformed to AML (N=29) | Poor-risk Cohort: Refractory/Relapsed AML, < 6 Mths Remission (N=46)
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 2 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 21 | 22 | 33
Hemoglobin (Blood and lymphatic system disorders) | 13 | 21 | 23
Lymphatics-Other (Blood and lymphatic system disorders) | 0 | 0 | 3
Left ventricular diastolic dysfunction (Cardiac disorders) | 2 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2 | 2
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 | 1 | 3
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 3 | 5 | 7
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Ocular/Visual-Other (Eye disorders) | 2 | 0 | 2
Pain - Eye (Eye disorders) | 0 | 2 | 3
Vision-blurred vision (Eye disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 10 | 6
Diarrhea (Gastrointestinal disorders) | 22 | 25 | 34
Distention/bloating, abdominal (Gastrointestinal disorders) | 1 | 9 | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 2 | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 | 1 | 5
Esophagitis (Gastrointestinal disorders) | 2 | 0 | 3
Gastrointestinal-Other (Gastrointestinal disorders) | 2 | 4 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 0 | 2 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 1 | 2 | 0
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4 | 5 | 4
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 20 | 22 | 24
Pain - Abdomen NOS (Gastrointestinal disorders) | 7 | 11 | 16
Pain - Oral cavity (Gastrointestinal disorders) | 1 | 0 | 7
Pain - Stomach (Gastrointestinal disorders) | 1 | 3 | 2
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 16 | 13 | 16
Constitutional Symptoms-Other (General disorders) | 0 | 3 | 3
Edema: head and neck (General disorders) | 1 | 4 | 1
Edema: limb (General disorders) | 5 | 14 | 8
Edema: viscera (General disorders) | 3 | 0 | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14 | 18 | 18
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 2 | 3 | 3
Injection site reaction/extravasation changes (General disorders) | 1 | 3 | 2
Pain - Chest/thorax NOS (General disorders) | 1 | 5 | 3
Pain - Pain NOS (General disorders) | 1 | 2 | 0
Pain-Other (General disorders) | 2 | 7 | 3
Rigors/chills (General disorders) | 3 | 10 | 8
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 3
Allergic reaction/hypersensitivity (Immune system disorders) | 4 | 3 | 1
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 | 2 | 6
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 5 | 5 | 10
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 5 | 3 | 6
Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums (Infections and infestations) | 3 | 1 | 2
Inf (clin/microbio) w/Gr 3-4 neuts - Skin (Infections and infestations) | 0 | 2 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Stomach (Infections and infestations) | 0 | 2 | 1
Infection-Other (Infections and infestations) | 2 | 4 | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 2 | 1 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 7 | 6 | 18
AST, SGOT (Investigations) | 5 | 10 | 18
Alkaline phosphatase (Investigations) | 4 | 8 | 9
Bilirubin (hyperbilirubinemia) (Investigations) | 8 | 7 | 13
Creatinine (Investigations) | 5 | 6 | 8
INR (of prothrombin time) (Investigations) | 0 | 4 | 6
Leukocytes (total WBC) (Investigations) | 16 | 16 | 18
Lymphopenia (Investigations) | 5 | 9 | 11
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 14 | 18 | 18
PTT (Partial thromboplastin time) (Investigations) | 1 | 0 | 9
Platelets (Investigations) | 18 | 19 | 20
Weight gain (Investigations) | 0 | 0 | 3
Weight loss (Investigations) | 4 | 3 | 8
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 | 20 | 19
Anorexia (Metabolism and nutrition disorders) | 4 | 14 | 10
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 9 | 19 | 16
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 | 11 | 14
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 | 6 | 6
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 | 10 | 12
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 | 11 | 15
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 | 4 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 12 | 20 | 24
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3 | 6 | 5
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 | 10 | 12
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 6 | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 7 | 8
Mental status (Nervous system disorders) | 3 | 0 | 1
Neurology-Other (Nervous system disorders) | 2 | 1 | 1
Neuropathy: sensory (Nervous system disorders) | 2 | 1 | 3
Ocular/Visual-Other (Nervous system disorders) | 2 | 0 | 2
Pain - Head/headache (Nervous system disorders) | 6 | 8 | 4
Taste alteration (dysgeusia) (Nervous system disorders) | 0 | 2 | 2
Confusion (Psychiatric disorders) | 1 | 3 | 4
Insomnia (Psychiatric disorders) | 3 | 5 | 6
Mood alteration - agitation (Psychiatric disorders) | 2 | 0 | 1
Mood alteration - anxiety (Psychiatric disorders) | 5 | 4 | 8
Mood alteration - depression (Psychiatric disorders) | 2 | 3 | 5
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 | 2 | 3
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 | 1 | 5
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 2 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 10
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 6
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 6
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 2 | 4 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 4
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 | 6 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 5 | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 | 15 | 11
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Flushing (Vascular disorders) | 0 | 2 | 4
Hemorrhage/Bleeding-Other (Vascular disorders) | 2 | 0 | 2
Hypertension (Vascular disorders) | 1 | 7 | 10
Hypotension (Vascular disorders) | 4 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT00840177/Prot_SAP_ICF_000.pdf